CLINICAL TRIAL: NCT05774197
Title: Leveraging mHealth to Deliver Integrated Pain-CBT, Opioid Monitoring, and Self-management Support for Advanced Cancer Patients Coping With Chronic Pain (STAMP+CBT)
Brief Title: Psychological Intervention Using Smartphone Technology to Alleviate Malignant Pain
Acronym: STAMP+CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STAMP+CBT; 1R21CA263838-01 (NIH)
Record Dates: First submitted 2023-02-15; First posted 2023-03-17 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Cancer Pain; Opioid Use; Cognitive Behavior Therapy
Keywords: STAMP (Smartphone Technology to Alleviate Malignant Pain); CBT (Cognitive Behavioral Therapy); mHealth (Mobile Health technology)
MeSH Terms: conditions — Cancer Pain; Color Vision Defects | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The STAMP+CBT application uses multi-media educational materials and survey algorithms assessing pain, medication usage, mood, stress, and sleep to improve pain management in this population. The primary objective is to determine the feasibility and acceptability during the 6-week study of the STAMP+CBT app (4-week intervention period and a 2-week post intervention period). Specifically, in this study 35 patients are enrolled and will be evaluated for their adherence to daily and weekly comprehensive symptom based self-assessments within the STAMP+CBT app.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STAMP+CBT app (Experimental): This app will allow the patient to access daily surveys designed to assess pain, stress, mood, and related symptoms.
  Based on patient-reported symptoms, this app will disseminate tailored education to manage the symptoms.
  Interventions: Behavioral: Cognitive Behavioral Therapy for pain

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for pain — Patient participating in this study will have survey assessments at baseline, 4 weeks (end of 4-week intervention period), and 6 weeks (end of 2-week post intervention period) assessing patient reported concerns, quality of life outcomes and usability of STAMP+CBT app. During this time, Patient will receive algorithm-based advice in response to their daily pain and mood surveys. These patients will be introduced to the extensive multi-media library of educational content covering medication support (e.g. using short and long-acting opioids, managing side effects, opioid safety); pain psychology (e.g. pain perception, pain and the stress response); health behaviors and pain (e.g. sleep hygiene); and skills training (e.g. activity pacing/ relaxation recordings).

SUMMARY:
The purpose of this study is to develop and pilot test a novel medical intervention (STAMP+CBT app) that will help patients track their pain, mood, opioid use and side effects while delivering tailored education and self-management advice for patients with advanced cancer.

DETAILED DESCRIPTION:
The primary purpose of this project is to determine the feasibility and acceptability of a novel mobile health application (STAMP+CBT app). The STAMP+CBT app (Smartphone Technology to Alleviate Malignant Pain + Cognitive Behavioral Therapy) seeks to provide education about pain medications alongside cognitive behavioral therapy techniques for pain to patients with advanced cancer. The application uses multi-media educational materials and survey algorithms assessing pain, medication usage, mood, stress, and sleep to improve pain management in this population. In this study, patients with advanced cancer at OU will participate in a single-arm, 6-week study of STAMP+CBT (4-week intervention period and a 2-week post-intervention period).

ELIGIBILITY:
Cohort Inclusion Criteria:

* Age ≥ 18 years
* Patient diagnosed with an active cancer diagnosis (locally advanced solid tumor malignancy, multiple myeloma, or other advanced hematologic malignancy), either undergoing active treatment or receiving treatment for an advanced cancer or are receiving supportive care
* Chronic pain related to cancer or treatment (> pain score of 4)
* Has an active prescription for at least one opioid medication to treat their cancer pain (i.e. not for post-surgical pain)
* Completed baseline survey

Cohort Exclusion Criteria:

* Patients in survivorship: patients who have completed their treatment regimens, are not actively receiving treatment for an advanced cancer, or have a cancer that is in remission
* Cognitive impairment that would interfere with study participation, as judged by treating clinician
* Inability to speak English (the intervention has not yet been translated to Spanish)
* Enrolled in hospice
* Currently hospitalized
* Use of transmucosal fentanyl, given safety concerns and ongoing risk mitigation program required to prescribe these (TIRF REMS)
* Pain primarily related to a recent surgery (within the last 2 weeks)

We will exclude adults who are unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant women, and prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desiree Azizoddin, PsyD, Principal Investigator — Stephenson Cancer Center
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 1 site from May 2023 to February 2024. The first patient was enrolled on May 4, 2023 and the last patient was enrolled on February 8, 2024.
Pre-assignment Details: Of 52 enrolled participants, 31 met inclusion criteria and assigned to the single arm study. Among 31 patients enrolled into the app, 16 completed all surveys.
Groups:
- STAMP+CBT App: This app will allow the patient to access daily surveys designed to assess pain, stress, mood, and related symptoms.
  Based on patient-reported symptoms, this app will disseminate tailored education to manage the symptoms.
  Cognitive Behavioral Therapy for pain: Patients participating in this study will have survey assessments at baseline, 4 weeks (end of 4-week intervention period), and 6 weeks (end of 2-week post intervention period) assessing patient reported concerns, quality of life outcomes and usability of STAMP+CBT app. During this time, Patient will receive algorithm-based advice in response to their daily pain and mood surveys. These patients will be introduced to the extensive multi-media library of educational content covering medication support (e.g. using short and long-acting opioids, managing side effects, opioid safety); pain psychology (e.g. pain perception, pain and the stress response); health behaviors and pain (e.g. sleep hygiene); and skills training (e.g. activity pacing/ relaxation recordings).
Period: Overall Study
Arm/Group | STAMP+CBT App
Started | 31
Completed | 16
Not Completed | 15
Not completed — Did not complete all the surveys required for study. | 15

BASELINE CHARACTERISTICS:
Groups:
- STAMP+CBT App: This app will allow the patient to access daily surveys designed to assess pain, stress, mood, and related symptoms.
  Based on patient-reported symptoms, this app will disseminate tailored education to manage the symptoms.
  Cognitive Behavioral Therapy for pain: Patient participating in this study will have survey assessments at baseline, 4 weeks (end of 4-week intervention period), and 6 weeks (end of 2-week post intervention period) assessing patient reported concerns, quality of life outcomes and usability of STAMP+CBT app. During this time, Patient will receive algorithm-based advice in response to their daily pain and mood surveys. These patients will be introduced to the extensive multi-media library of educational content covering medication support (e.g. using short and long-acting opioids, managing side effects, opioid safety); pain psychology (e.g. pain perception, pain and the stress response); health behaviors and pain (e.g. sleep hygiene); and skills training (e.g. activity pacing/ relaxation recordings).
Arm/Group | STAMP+CBT App
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.41 (12.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Rural Dwelling [Count of Participants; unit: Participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Complete More Than 2/3rd of the Study Modules at the End of 4 Weeks of Intervention to Determine Feasibility of the STAMP+CBT App
Description: Patients will be assigned surveys at baseline, 4-week intervention period and 2 weeks post intervention period (6 weeks from baseline). Based on that patient's overall adherence rate/app retention rates will be calculated and intervention will be considered feasible if more than 70% of subjects complete any activity on the app at least 50% of days on study.
Time Frame: 4-weeks
Population: Patients who enrolled in the study and used the app
Measure: Count of Participants; unit: Participants
Arm/Group | STAMP+CBT App
Number analyzed (Participants) | 31
Participants | 19

2. Primary Outcome: Proportion of Patients Who Rate the Acceptability Items 4 or Higher on the App.
Description: Patients will be assigned surveys at baseline, 4-week intervention period and 2 weeks post intervention period (6 weeks from baseline). In response to the survey's patient will be assigned tailored psychological intervention for advanced cancer pain. During the trial, these interventions will be considered acceptable only if 80% or more of the acceptability items are rated 4 or higher/5; Lower rating will lead to app refinements.
Time Frame: 6-weeks
Population: Patients who enrolled in the study and used the app and completed the survey
Measure: Count of Participants; unit: Participants
Arm/Group | STAMP+CBT App
Number analyzed (Participants) | 21
Participants | 15

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | STAMP+CBT App
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-23): https://cdn.clinicaltrials.gov/large-docs/97/NCT05774197/Prot_SAP_000.pdf